CLINICAL TRIAL: NCT07100964
Title: The Effect of Multiple Oral Doses of Carbamazepine on the Single-oral-dose Pharmacokinetics of Nerandomilast in Healthy Male Trial Participants (an Open-label, Two-treatment, Two- Period Fixed Sequence Trial)
Brief Title: A Study in Healthy Men to Test Whether Carbamazepine Influences the Amount of Nerandomilast in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0119; 2025-521279-30-00 (Registry Identifier: CTIS); U1111-1320-6353 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nerandomilast alone followed by nerandomilast + carbamazepine (Experimental)
  Interventions: Drug: nerandomilast; Drug: carbamazepine

INTERVENTIONS:
Drug: nerandomilast — nerandomilast
  Other Names: JASCAYD®
Drug: carbamazepine — carbamazepine

SUMMARY:
The main objective of this trial is to investigate the effect of carbamazepine on pharmacokinetics of nerandomilast.

ELIGIBILITY:
Inclusion Criteria :

1. Healthy male trial participant according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), body weight, 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body Mass Index (BMI) of 18.5 to 29.9 kg/ m^2 (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
5. If sexually active, sexual abstinence or use of a condom for at least 2 weeks after the last administration of carbamazepine.

Exclusion Criteria :

1. Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or ECG, neurological examination and skin inspection) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate (PR) outside the range of 50 to 90 bpm
3. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
4. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, haematological, neurological, psychiatric or hormonal disorders assessed as clinically relevant by the investigator
5. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
6. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders including but not limited to depression and suicidal behaviour
7. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-08-11 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz) | Up to 30 days
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 30 days

SECONDARY OUTCOMES:
Area under the Plasma Concentration Curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC 0-∞) | Up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com